CLINICAL TRIAL: NCT04593953
Title: Efficacy of Thoraco-Lumbar Interfascial Plane (TLIP) Block for Postoperative Analgesia of Lumbar Spinal Fusion
Brief Title: Efficacy of TLIP Block for Postoperative Analgesia of Lumbar Spinal Fusion
Acronym: ETLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2020/01
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Lumbar Spinal Fusion
Keywords: TLIP block; Lumbar spinal fusion; Regional anesthesia; Ropivacaine; Postoperative analgesia; Ultrasound; Pain management; Opioids
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: To minimize assessment bias, patients and evaluators (nurse and physiotherapist) will be unaware of the intervention group. Only the investigator, who will include the patient and will realize the procedure, will know the arm of randomization.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL (No Intervention): Standard general anesthesia
- TLIP (Experimental): Standard general anesthesia + TLIP block
  Interventions: Procedure: TLIP

INTERVENTIONS:
Procedure: TLIP — Injection of 40 ml of ropivacaine 0.25% (2 injections of 20 ml on each side) between multifidus and longissimus muscles.
  Arms: TLIP

SUMMARY:
Spinal surgery is associated with severe pain in the immediate postoperative period. In a recent study evaluating pain intensity on the first day after surgery in a large range of surgical procedures, among the six most painful surgeries, three were major spinal procedures. Spinal surgery causes an accumulation of several types of pain. Incisional pain results from activation of peripheral nociceptors. Musculoskeletal pain arises from damage to structures, such as bone, ligaments, muscles, intervertebral disks, and zygapophyseal joints. In addition, neuropathic pain arises from compression and damage to nerve roots exiting the spinal canal and sometimes damage to the spinal cord itself.

Postoperative pain management requires multimodal analgesia, combining drugs and injection of a local anesthetic (LA) in order to reduce opioid consumption after surgery. Among regional anesthesia (RA) techniques, the thoraco-lumbar interfascial plane block (TLIP) was considered. It offers an effective and safe analgesia during the first 24h after herniated lumbar disc surgery. Ultrasound-guided TLIP block involves injection of LAs between longissimus and multifidus muscles (spinal lombar muscles). This injection allows to block the dorsal rami of spinal nerves innervating the paravertebral muscles and the vertebrae.

The objective of this study is to evaluate the interest of TLIP block to improve the postoperative analgesia in patients undergoing lumbar spinal fusion surgery.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind (participant and care provider assessing outcomes), parallel-group controlled, trial assessing the interest of the association of TLIP block to general anesthesia for postoperative analgesia management in patients undergoing posterior lumbar spinal fusion.

This study compares two groups:

"Control" group: standard general anesthesia. "TLIP" group: standard general anesthesia + TLIP block with an injection of 40 ml of ropivacaine 0.25% (2 injections of 20 ml on each side) between multifidus and longissimus muscles.

• General anesthesia

General anesthesia will be standardized in the two groups:

* Induction with propofol 2-3 mg/kg, sufentanyl 0.2-0.3 µg/kg and ketamine 0.3 mg/kg
* Intubation facilitated according centre's protocol and ventilation performed with 50% oxygen and 50% air in order to maintain normocapnia and normoxia.
* Anesthesia maintained according to the centre's usual care.
* Prevention of postoperative nausea and vomiting (NVPO) according centre's protocol.

  * TLIP block technique ("TLIP" group only) The regional anesthesia procedure will be performed under general anesthesia and will be guided by ultrasound with high-frequency linear probe, patient in prone position or genupectoral (knee-chest) position. The probe will be positioned in order to have an axial view of lumbar vertebrae. The 3rd lumbar vertebra (L3), the 4th lumbar vertebra (L4) and the 5th lumbar vertebra (L5) will be identified after initial identification of the sacrum. A needle will be inserted in plane (IP) and advanced to reach the interspace between the multifidus and the longissimus muscles on the tip of the articular process. For each patient, the block will be performed bilaterally by injecting of 20 ml of Ropivacaine 0.25% on each side. Before each procedure, a skin disinfection will be carried out using an alcoholic iodine solution.

Patients will not receive any LA by intravenous injection or infiltration.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old,
* Undergoing posterior lumbar spinal one-level or two-level fusion surgery (L3-L4, L4-L5 and/or L5-S1),
* Having signed a written informed consent form,
* Affiliation to the social security system.

Exclusion Criteria:

* Contraindication for regional anesthesia (allergy to local anesthetics, neuropathic disease, infection at the puncture site, coagulation disorder, refusal of the technique,…)
* Contraindication to nonsteroidal anti-inflammatory drugs,
* Patient who have already had a spinal surgery,
* Patient with chronic pain syndrome (use > 3 months of morphine, opioid analgesics of class 3, pregabalin or gabapentin) or fibromyalgia,
* A mental or linguistic inability to understand the study,
* Patient under protection of the adults (guardianship, curators or safeguard of justice),
* Pregnant or or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Morphine consumption in the first 24 hours post-surgery | 24 hours
  Total amount of morphine (mg) administered during the first 24 hours post-surgery. The reference time t0 will be the time of skin incision.

SECONDARY OUTCOMES:
Morphine consumption in the first 48 hours post-surgery | 48 hours
  Total amount of morphine (mg) administered during the first 48 hours post-surgery
Morphine consumption in the post-anesthesia care unit (PACU) | 6 hours
  Total amount of morphine (mg) administered in PACU
Duration of postoperative analgesia | 48 hours
  Time (in minutes) between the skin incision (t0) and the first administration of morphine in PACU or in ward.
Postoperative pain: Visual Analogue Scale (VAS) | 48 hours
  Pain scores using a Visual Analogue Scale (VAS) ranging from 0 to 10 (0= no pain; 10= worst imaginable pain). These scores will be recorded before surgery, in PACU and four times a day (morning, afternoon, evening and night) during the first 48 hours post-surgery, both at rest and during exercises (walk with the physiotherapist).
Postoperative quality of recovery | 72 hours
  15-item Quality of Recovery (QoR-15) scale ranging from 0 to 10 (0= very poor recovery; 150= excellent recovery). This multidimensional questionnaire assesses five domains of patient-reported health status: pain, physical comfort, physical independence, psychological support and emotional state.
Side effects associated with opioids | 72 hours
  Incidence of side effects associated with morphine: nausea and vomiting, drowsiness, acute urinary retention.
Rate of complications | 20 minutes, 72 hours
  Poor distribution of local anesthetic and rhythm disorders linked to an intravascular injection assessed during regional anesthesia procedure and during the 20 minutes following the block.
  Infection at the injection site and mechanical complications: hematoma, assessed 72h post-surgery.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Privé Jean Mermoz, Lyon
  - CMC Ambroise Paré, Neuilly-sur-Seine, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No